CLINICAL TRIAL: NCT05195645
Title: AbataCept for the Treatment of Immune-cHeckpoint Inhibitors Induced mYocarditiS
Acronym: ACHLYS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP210303
Record Dates: First submitted 2021-12-10; First posted 2022-01-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Myocarditis
Keywords: Myocarditis; Immune-checkpoint-inhibitors (ICI); ICI-induced myocarditis; immune-related adverse events; Abatacept; Dose-finding
MeSH Terms: conditions — Myocarditis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A-10mg/kg (Experimental): Patients in arm A will receive doses of 10 mg/kg of Abatacept
  Interventions: Drug: Abatacept 250 MG
- B-20mg/kg (Experimental): Patients in arm B will receive doses of 20 mg/kg of Abatacept
  Interventions: Drug: Abatacept 250 MG
- C-25mg/kg (Experimental): Patients in arm C will receive doses of 25 mg/kg of Abatacept
  Interventions: Drug: Abatacept 250 MG

INTERVENTIONS:
Drug: Abatacept 250 MG — Abatacept will be administered by intravenous injection over 1h15 to 2h30 on D1, D5+/-2 and D14+/-2 at 10mg/kg (arm A), or 20mg/kg (arm B) or 25mg/kg (arm C) depending on the randomization (max 3 000 mg per administration). Starting Day 21 (after evaluation of the primary outcome), other injection of abatacept may be given (D22 at D90) with dosage (10 or 20mg/kg max) decided by the treating physician (max 2 500 mg per administration) as a function of the relapse or not of the ICI myocarditis after immunosuppressant therapeutics tapering. After day 21, the administrations will be carried out in open but the blind administration 1 to 3 (D1 to D21) will be kept.
  Other Names: ORENCIA® BMS

SUMMARY:
Immune-checkpoint-inhibitors (ICI) have revolutionized treatment for about 20 cancer types. They unleash anti-tumor immune responses. Unfortunately, in 0.36-1.23% of patients, this activation can also lead to lethal immune-related adverse events (irAEs) that can affect any organ. Among those irAEs, ICI-induced myocarditis was the most frequently fatal with death rate reaching 50% in a large case-series of over 100 patients.

This study is a dose-finding Phase II trial where 3 abatacept IV regimen (A-10 mg/kg; B-20 mg/kg and C-25 mg/kg at Day0, Day5+/-2, Day14+/-2) will be tested aiming at reaching promptly (after the first dose) and sustainably a CD86RO≥80% during the first 3 weeks of ICI-myocarditis management. The main objective is to find the lowest dose required to achieve a circulating monocytes CD86RO≥80% within the first week of treatment and sustainably over three weeks. The target population is all adult patients with cancer (all cancer types) treated by immune checkpoint inhibitors (anti-PD1, anti-PDL1, anti-CTLA4 monotherapies or combination) and presenting drug-induced myocarditis.

DETAILED DESCRIPTION:
Immune-checkpoint-inhibitors (ICI) have revolutionized treatment for about 20 cancer types. They unleash anti-tumor immune responses. Unfortunately, in 0.36-1.23% of patients, this activation can also lead to lethal immune-related adverse events (irAEs) that can affect any organ. Among those irAEs, ICI-induced myocarditis was the most frequently fatal with death rate reaching 50% in a large case-series of over 100 patients. Other severe irAEs are pneumonitis, hepatitis and neuromyotoxicities (myositis, myasthenia gravis-like syndrome) with death rates of 20-25%. Co-occurrence of irAEs affecting multiple organs is frequent (30% for myocarditis and myositis) as they share underlying mechanisms with macrophages and cytotoxic T-cell infiltrates leading to organ destruction.

While rigorous studies for the treatment of irAEs are lacking, consensus guidelines recommend treatment with high-dose corticosteroids with progressive tapering and withholding ICI. When symptoms and biological markers do not improve, other immunosuppressive drugs (mycophenolate-mofetil, methotrexate, cyclosporine, cyclophosphamide, azathioprine, antithymocyte globulin, infliximab, tocilizumab, and rituximab) can be considered, depending on organs affected. Intravenous immunoglobulin or plasmapheresis can also be considered. In patients developing myocarditis, available therapeutics produce poor results and the fatality rate (40-50%) has stagnated between 2014-2019 despite increasing glucocorticoids use. No treatment has been shown to improve this situation. Thus, better reversal agents' strategies are urgently needed in the context of the increasing use of ICI and of associated irAEs. Abatacept and belatacept (CTLA4-immunoglobulin fusion proteins) have very promising properties: they inhibit CD80/CD86 mediated T-cell co-stimulation at the level of dendritic-cells, thereby abrogating activation of the T-cells upstream of the CTLA4 and PD1/PDL1 pathways. "CTLA4 agonists" leads to global T-cell anergy with limited off-target effects, and specifically reverse ICI-activated pathways.

Abatacept is currently indicated in rheumatological disorders such as rheumatoid arthritis and belatacept is indicated in kidney rejection transplantation prophylaxis. In these latter indications, the circulating monocytes CD86 receptor occupancy (CD86RO) by "CTLA4 agonists" is a relevant pharmacodynamic biomarker of their clinical activity. The target CD86RO cut-off should be over 80%.

Confirming the rationale for "CTLA4 agonists" use in ICI-myocarditis, the investigators recently showed that abatacept was able to alleviate fatal myocarditis in CTLA4/PD1 genetic knock-out mice model. Finally, this group recently described the first cases of glucocorticoid-refractory myocarditis induced by nivolumab (anti-PD1) which resolved after treatment with abatacept. This success prompted the investigators to treat over 15 ICI-myocarditis patients in their institution and several other teams to use abatacept in ICI-induced myocarditis with encouraging results. Though, in their experience, initial doses of abatacept needed to promptly reach CD86RO≥80% in ICI-myocarditis setting were much higher than those needed in its usual indications. Due to abatacept slow time to onset, combination with ruxolitinib (a JAK inhibitor) on top of corticosteroids was also proposed in ICI myocarditis management with very promising results (ICI-myotoxicity related mortality dropped from 60% on corticosteroids + 2nd line abatacept to 3% in 1st line abatacept + ruxolitinib + corticosteroids (https://doi.org/10.1158/2159-8290.CD-22-1180).

This study is a dose-finding Phase II trial where 3 abatacept IV regimen (A-10 mg/kg; B-20 mg/kg and C-25 mg/kg at Day0, Day5+/-2, Day14+/-2) will be tested aiming at reaching promptly (after the first dose) and sustainably a CD86RO≥80% during the first 3 weeks of ICI-myocarditis management. The main objective is to find the lowest dose required to achieve a circulating monocytes CD86RO≥80% within the first week of treatment and sustainably over three weeks. The target population is all adult patients with cancer (all cancer types) treated by immune checkpoint inhibitors (anti-PD1, anti-PDL1, anti-CTLA4 monotherapies or combination) and presenting drug-induced myocarditis.

Abatacept will be added to the standard of care of these severe ICI myocarditis patients, which include preferentially prednisone and ruxolitinib, tapered as a function of the bio-clinical evolution of ICI-myocarditis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Weight ≥ 40 kg and ≤ 125 kg
3. Patients treated with ICI immunotherapy (monotherapy or combination), including anti-PD1, anti-PDL1, anti-CTLA4; and including any type of cancer (even those in which ICI is not currently approved by regulatory)
4. Definite, probable or possible ICI-induced myocarditis according to the diagnostic criteria of the most recent expert consensus recommendations (e.g27, to be updated with any new recommendations to be published)
5. Severe or corticosteroid-resistant ICI-myocarditis:

   * Severe ICI-myocarditis is defined either 1/ by the appearance of an alteration of the LVEF<50% or a wall motion kinetics abnormality, or 2/ by the appearance of ventricular tachycardias or high-grade conductive disorders (atrioventricular block grade 2 or 3) or 3/ by the association with myasthenia gravis-like-syndrome (diplopia, ptosis, diaphragmatic dysfunction, dysarthria, dysphonia, dysphagia) or 4/ by troponin-T levels above 32 times the upper limit of the normal (a population at very high-risk ~75% of major cardiomuscular events in the month following initial presentation, cf. Circulation. 2023 Aug 8;148(6):473-486).
   * Corticosteroid-resistant ICI-myocarditis is defined by the absence of decrease in troponin levels or the appearance/persistence of severity criteria despite receiving prednisone dose ≥0.5 mg/kg/day for ≥2 days.
6. Signature of informed consent before any trial procedure from the patient or legal representative or the close relative
7. Patients covered by social security regimen (excepting AME)
8. Withhold of ICI

Exclusion Criteria:

1. Untreated and/or uncontrolled bacterial, fungal, or viral infection
2. Pregnancy, breast-feeding or planning to become pregnant during the study period
3. For women of childbearing age, lack of effective contraception throughout the duration of participation in the study
4. Being treated with abatacept or belatacept within 3 months prior to inclusion
5. Known hypersensitivity to abatacept or belatacept
6. Being treated with anti-thymoglobulin, or alemtuzumab within 6 weeks of the first scheduled dose of abatacept
7. Patient participating to another interventional study (RIPH 1 only)
8. People under legal protection measure (tutorship, curatorship or safeguard measures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an adequate circulating monocytes CD86 receptor occupancy (CD86RO) saturation ≥ 80% | CD86RO will be assessed versus baseline levels (1 to 3 hours before 1st abatacept administration for baseline) and then, once 1 to 3 hours and 12 to 72 hours after the 1st, 2nd and 3rd abatacept administration, and at Day 21 .
  A patient will be considered with an adequate CD86RO saturation (≥80%) within the first weeks of treatment if at least three CD86RO assessment are over 80% until Day 21 after the first abatacept administration.

SECONDARY OUTCOMES:
Quantification of proxies reflecting the resolution of systemic immune activation | one to 3 hours before abatacept treatment (Baseline), once 1 to 3 hours after, and once 12 to 72 hours after the first administration, 2nd and 3rd abatacept dose, then every ten days up to day 90, and then every three months up to a year of follow-up
  % of regulator T-cells CTLA4+ will be assessed versus baseline levels (one to 3 hours before abatacept treatment, preferentially before corticosteroids or any other immunossupressant intake). In case of additional doses of abatacept, it will also be additionally measured one to 3 hours before and one to three hours after each dose of abatacept.
Quantification of proxies reflecting the resolution of systemic immune activation | one to 3 hours before abatacept treatment (Baseline), once 1 to 3 hours after, and once 12 to 72 hours after the first administration, 2nd and 3rd abatacept dose, then every ten days up to day 90, and then every three months up to a year of follow-up
  Levels of pro and anti-inflammatory cytokines will be assessed versus baseline levels (one to 3 hours before abatacept treatment, preferentially before corticosteroids or any other immunossupressant intake). In case of additional doses of abatacept, it will also be additionally measured one to 3 hours before and one to three hours after each dose of abatacept.
Quantification of proxies reflecting the resolution of systemic immune activation | one to 3 hours before abatacept treatment (Baseline), once 1 to 3 hours after, and once 12 to 72 hours after the first administration, 2nd and 3rd abatacept dose, then every ten days up to day 90, and then every three months up to a year of follow-up
  C-reactive protein levels will be assessed versus baseline levels (one to 3 hours before abatacept treatment, preferentially before corticosteroids or any other immunossupressant intake). In case of additional doses of abatacept, it will also be additionally measured one to 3 hours before and one to three hours after each dose of abatacept.
Quantification of proxies reflecting the resolution of systemic immune activation | one to 3 hours before abatacept treatment (Baseline), once 1 to 3 hours after, and once 12 to 72 hours after the first administration, 2nd and 3rd abatacept dose, then every ten days up to day 90, and then every three months up to a year of follow-up
  % of circulating T-cells expressing PDL1 will be assessed versus baseline levels (one to 3 hours before abatacept treatment, preferentially before corticosteroids or any other immunossupressant intake). In case of additional doses of abatacept, it will also be additionally measured one to 3 hours before and one to three hours after each dose of abatacept.
Quantification of proxies reflecting the resolution of systemic immune activation | one to 3 hours before abatacept treatment (Baseline), once 1 to 3 hours after, and once 12 to 72 hours after the first administration, 2nd and 3rd abatacept dose, then every ten days up to day 90, and then every three months up to a year of follow-up
  % of circulating T-cells expressing PD1 will be assessed versus baseline levels (one to 3 hours before abatacept treatment, preferentially before corticosteroids or any other immunossupressant intake). In case of additional doses of abatacept, it will also be additionally measured one to 3 hours before and one to three hours after each dose of abatacept.
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 90
  Quantification of the corticosteroid decrease kinetics (total cumulative dose)
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 21
  Quantification of the corticosteroid decrease kinetics (total cumulative dose)
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 90
  Quantification of the corticosteroid decrease kinetics (time to weaning)
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 21
  Quantification of the corticosteroid decrease kinetics (time to weaning)
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 90
  Quantification of the proportion of patients for whom it was necessary to add other immunosuppressants in addition to glucocorticoids to control the disease
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 21
  Quantification of the proportion of patients for whom it was necessary to add other immunosuppressants in addition to glucocorticoids to control the disease
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 90
  Cumulative dose of other immunosuppressants added to glucocorticoids in patients for whom it was necessary to add this immunossupressant to control the disease
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 21
  Cumulative dose of other immunosuppressants added to glucocorticoids in patients for whom it was necessary to add this immunossupressant to control the disease
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 90
  Time to weaning of other immunosuppressants added to glucocorticoids in patients for whom it was necessary to add this immunossupressant to control the disease
Quantification of proxies reflecting the resolution of systemic immune activation | Between Day 0 and Day 21
  Time to weaning of other immunosuppressants added to glucocorticoids in patients for whom it was necessary to add this immunossupressant to control the disease
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Incidence of heart failure (defined as left-ventricular drop below 50%)
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Incidence of life-threatening cardiac arrhythmias (defined a sustained >30 seconds ventricular tachycardia epidose, ventricular fibrillation, cardiac arrest, sinus arrest >4 seconds and complete atrio-ventricular block).
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Evolution of grading of the cardiomyotoxicity overall
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Evolution of grading of the cardiomyotoxic sub-features (cardiac dysfunction)
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Evolution of grading of the cardiomyotoxic sub-features (cardiac pro-arrhythmias)
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Evolution of grading of the cardiomyotoxic sub-features (respiratory muscle dysfunction)
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Evolution of grading of the cardiomyotoxic sub-features (dysphagia)
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  troponin-T and -I maximal value
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Area under the curve of troponin levels
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Area under the curve of Creatine Kinase level
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Creatine Kinase level maximal value
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  NT-proBNP maximal value
Quantification of proxies reflecting the resolution of myocarditis | Between Day 0 and Day 21, and Day 90
  Area under the curve of NT-proBNP
Quantification of proxies reflecting the resolution of myocarditis | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  left ventricular ejection fraction by echocardiography
Quantification of proxies reflecting the resolution of myocarditis | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Cardiac inflammation and myocardial edema quantification by cardiac MRI
Quantification of proxies reflecting the resolution of myocarditis | At admission, Day 5, Day 14, Day 21, Day 90 and then every 3 months up to one year
  Arrhythmias and ventricular conductive disorders quantified on 48hours electrocardiographic Holter acquisitions
Quantification of proxies reflecting the resolution of myocarditis | At admission, Day 21, Day 90, 6 months and one year
  Humoral autoimmunity against the myocardium or the muscles (anti- cardiac troponin I and T, anti-titin, anti-muscle specific kinases (musK), anti-acetylcholine receptor antibodies).
Quantification of proxies reflecting the involvement and resolution of any associated myositis | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Presence/absence on electromyogram assessment of : myogenic syndrome (0/1), diaphragmatic nerve dysfunction (0/1), decrement on assessment of neuromuscular dysfunction (0/1)
Quantification of proxies reflecting the involvement and resolution of any associated myositis: | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Number of significant hypoxemic episodes by capnography
Quantification of proxies reflecting the involvement and resolution of any associated myositis | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Proportion of time with abnormal CO2 (%) by capnography.
Quantification of proxies reflecting the involvement and resolution of any associated myositis | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Maximum C02 (mmHg) by capnography
Quantification of proxies reflecting the involvement and resolution of any associated myositis | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Presence/absence of restrictive syndrome (0/1) by functional respiratory exploration.
  Presence/absence of sign of diaphragmatic failure (0/1) by functional respiratory exploration.
Quantification of proxies reflecting the involvement and resolution of any associated myositis | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Maximal/minimal Inspiratory Pressure (mmHg) by functional respiratory exploration.
Quantification of proxies reflecting the involvement and resolution of any associated myositis: | These modalities will be assessed at least once as soon as possible after admission, 3 months and one year after the first abatacept administration.
  Excursion of the right and left diaphragmatic border (mm) by diaphragmatic MRI and echography
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | Throughout the study completion (up to one year after randomization)
  Determination of the volume of distribution (Liter) by using all the evaluated abatacept circulating levels
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | Throughout the study completion (up to one year after randomization)
  Determination of the terminal half-life (days) by using all the evaluated abatacept circulating levels
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | Throughout the study completion (up to one year after randomization)
  Determination of clearance (ml/min/kg) by using all the evaluated abatacept circulating levels
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | Throughout the study completion (up to one year after randomization)
  Determination of maximum concentration of circulating abatacept (Cmax, µg/ml) by using all the evaluated abatacept circulating levels
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | Throughout the study completion (up to one year after randomization)
  Determination of residual concentration of circulating abatacept (Cmin, µg/ml) by using all the evaluated abatacept circulating levels
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | Throughout the study completion (up to one year after randomization)
  Determination of time to Cmax (hours) by using all the evaluated abatacept circulating levels
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | Abatacept, CD86RO and troponin-T blood levels assessed minimum at baseline (1-3h before abatacept) and once 1-3h after, and 12-72h after 1st, 2nd, 3rd and extra abatacept doses, then every 10days up to day90, and then every 3months up to 1year.
  Modelling of the 50% median effective concentration (µg/ml) of abatacept to saturate CD86 receptor on circulating monocytes (%) and to achieve troponin safety levels targets
Pharmacokinetic/pharmacodynamic (PK-PD) modelling of abatacept in ICI-myocarditis | ADA will be searched at inclusion (before 1st abatacept intake), and then at day 21, 3 months and 6 months after randomization
  Presence of Abatacept anti-drug antibody (ADA, 0/1)
Quantification of tumor progression | The imaging modalities will be assessed at least once as soon as possible after admission, after 3 months and one year after abatacept start.
  Quantification of tumor progression by appropriate examination depending on the tumor type (e.g. CT-scan for lung or renal cancer) using the best monitoring work-up used in standard of care.
Quantification of tumor progression | Progression free survival rate at 90days, 6 months and 12 months
  Progression free survival defined as time from randomization to progression according to RECIST criteria
Quantification of the number and severity (in particular fatal) of adverse events, in particular infectious, according to the CTCAE v5.0 classification. | Full clinical examination : Before starting treatment, during the treatment course and during 1 year / Active clinical monitoring during the treatment course and for 1 year / Biological monitoring : During the first 4 weeks, at 3 months and one year
  A Full clinical examination searching for any ongoing infection before starting treatment and active clinical monitoring of any sign of new infection during the treatment course and for 1 year.
  The biological monitoring will include with a blood PCR seeking for CMV reactivation weekly for 4 weeks and then at 3 months and one year (in patients carrying a positive serology for CMV); as well as a blood next generation sequencing seeking for pathogens will be assessed at least once as soon as possible after admission, then at day 14, 3 months and one year after the first abatacept administration.
Overall survival | Between Day 0 and 1 month, 3 months, 6 months and 12 months
  Proportion of patients alive without myotoxicity grade >2
Overall survival | Between Day 0, and 3 months, 6 months and 12 months
  Proportion of patients alive

CONTACTS AND LOCATIONS:
Overall Officials: Joe-Elie SALEM, Pr, Study Director — Pitie Salpetriere Hospital , APHP
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Salem JE, Ederhy S, Belin L, Zahr N, Tubach F, Procureur A, Allenbach Y, Rosenzwjag M, Bretagne M. Abatacept dose-finding phase II triaL for immune checkpoint inhibitors myocarditis (ACHLYS) trial design. Arch Cardiovasc Dis. 2025 Feb;118(2):106-115. doi: 10.1016/j.acvd.2024.12.005. Epub 2024 Dec 20. PMID 39743436